CLINICAL TRIAL: NCT00686426
Title: Role of Dairy Products in Weight Maintenance: Prevention of Weight Regain Following Weight Loss
Brief Title: Role of Dairy Products in Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Dairy Council (Other); University of Kansas (Other)
Responsible Party: Michael B. Zemel, the University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DMI-993
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Obesity; Weight Gain
Keywords: Obesity; Weight gain; regain; dairy; calcium
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Low Dairy
  Interventions: Dietary Supplement: Dairy Foods
- 2 (Experimental): Adequate Dairy
  Interventions: Dietary Supplement: Dairy Foods

INTERVENTIONS:
Dietary Supplement: Dairy Foods — Adequate dairy (> 3 standard daily servings)
  Arms: 2
Dietary Supplement: Dairy Foods — < 1 standard dairy serving/day
  Arms: 1

SUMMARY:
The goal of the current study is to determine the role of dairy in similarly preventing weight and fat re-gain in obese adults who have successfully completed a weight loss diet program.240 obese subjects will undergo a meal-replacement-based weight loss plan designed to produce a 10 kg weight loss in 8-12 weeks. Upon achieving the weight loss goal, subjects will be randomly assigned to either a low-dairy or high-dairy eucaloric weight maintenance diet for two years. Macronutrient distribution will be maintained constant and set at approximately the U.S. average. Primary outcomes include changes in body weight, body fat and anatomical distribution of fat (via dual x-ray absorptiometry) and resting metabolic rate and substrate oxidation (via respiratory calorimetry); Secondary outcomes include blood pressure, circulating glucose, insulin, lipids and calcitrophic hormones. on prevention of weight regain in humans has not yet been assessed in clinical trials.

DETAILED DESCRIPTION:
Dietary calcium plays a pivotal role in the regulation of energy metabolism, as we have found high calcium diets to attenuate adipocyte lipid accretion and weight gain during periods of over-consumption of an energy-dense diet and to increase lipolysis and preserve thermogenesis during caloric restriction, thereby markedly accelerating weight loss. Our studies of the agouti gene demonstrate a key role for intracellular Ca2+ in regulating adipocyte lipid metabolism and triglyceride storage, with increased intracellular Ca2+ resulting in stimulation of lipogenic gene expression and lipogenesis and suppression of lipolysis, resulting in adipocyte lipid filling and increased adiposity. Moreover, the increased calcitriol produced in response to low calcium diets stimulates adipocyte Ca2+ influx and, consequently, promotes adiposity, while higher calcium diets inhibit lipogenesis, promote lipolysis, lipid oxidation and thermogenesis and inhibit diet-induced obesity in mice. Notably, dairy sources of calcium exert markedly greater effects in attenuating weight and fat gain and accelerating fat loss. This augmented effect of dairy products versus supplemental calcium is likely due to additional bioactive compounds in dairy which act synergistically with calcium to attenuate adiposity. These concepts are confirmed by both epidemiological and clinical data which demonstrates that increasing dietary calcium results in significant reductions in adipose tissue mass in obese humans in the absence of caloric restriction and markedly accelerates the weight and body fat loss secondary to caloric restriction, while dairy products exert markedly greater (nearly two-fold compared to calcium supplements) effects. These data indicate an important role for dairy products in both the prevention and treatment of obesity. However, weight maintenance following successful weight loss (i.e. prevention of regain) is at least as important as strategies to initially achieve weight loss, as most individuals who successfully lose weight are not successful in maintaining this weight loss. We have recently demonstrated that ad libitum re-feeding of dairy-rich following weight loss in mice on an energy restricted mice prevented the suppression of adipose tissue lipolysis and fat oxidation that otherwise accompanies such re-feeding and markedly upregulated skeletal muscle fat oxidation. Consequently, although animals re-fed low calcium diets rapidly regained all of the weight and fat that had been lost, animals fed high calcium diets exhibited a shift in energy partitioning and a 50-85% reduction in weight and fat gain; moreover, dairy exerted markedly greater effects than supplemental calcium on weight and fat regain. However, the effect of dairy on prevention of weight regain in humans has not yet been assessed in clinical trials. Accordingly, the goal of the current study is to determine the role of dairy in similarly preventing weight and fat re-gain in obese adults who have successfully completed a weight loss diet program.

340 obese subjects will undergo a meal-replacement-based weight loss plan designed to produce a 10 kg weight loss in 8-12 weeks. Upon achieving the weight loss goal, subjects will be randomly assigned to either a low-dairy or high-dairy eucaloric weight maintenance diet for two years. Macronutrient distribution will be maintained constant and set at approximately the U.S. average. Primary outcomes include changes in body weight, body fat and anatomical distribution of fat (via dual x-ray absorptiometry) and resting metabolic rate and substrate oxidation (via respiratory calorimetry); Secondary outcomes include blood pressure, circulating glucose, insulin, lipids and calcitrophic hormones.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 30-39.9 kg/m2
* Age 25-50 years
* No more than 3 kg weight loss during past three months
* Negative pregnancy test at entry; women of childbearing potential may be enrolled if they have had a tubal ligation or use one of the following means of contraception: condom, diaphragm, oral or implanted contraceptives, or intrauterine device. Women in exclusive relationships with male partners who have had a successful vasectomy will not be required to use any additional means of birth control.

Exclusion Criteria:

* BMI < 30 or >40
* Type II diabetes requiring the use of any oral antidiabetic agent and/or insulin (because of confounding effects on body weight regulation)
* Adverse response to study foods (lactose intolerance, dairy intolerance, dairy allergy); this will be determined by self-report.
* History or presence of significant metabolic disease which could impact on the results of the study (i.e. endocrine, hepatic, renal disease)
* History of eating disorder
* Presence of active gastrointestinal disorders such as malabsorption syndromes
* Pregnancy or lactation
* Use of obesity pharmacotherapeutic agents within the last 6 months
* Use of over-the-counter anti-obesity agents (e.g. those containing phenylpropanalamine, ephedrine and/or caffeine) within the last 6 months
* Recent (past 12 weeks) use of tobacco
* Recent (current or past 12 weeks) use of any psychotropic medication
* Recent (past four weeks) initiation of an exercise program
* Recent (past twelve weeks) initiation of hormone replacement therapy or change in HRT regimen
* Recent (past twelve weeks) initiation of hormonal birth control or change in hormonal birth control regimen

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 338 (Actual)
Dates: Start 2003-11; Primary Completion 2007-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Body weight change | 6 months
Body Fat Change | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zemel, PhD, Principal Investigator — University of Tennessee; Joseph E Donnelly, PhD, Principal Investigator — University of Kansas
Locations (2):
- United States (2):
  - University of Kansas, Lawrence, Kansas
  - The University of Tennessee, Knoxville, Tennessee

REFERENCES:
- [Derived] Zemel MB, Sun X, Sobhani T, Wilson B. Effects of dairy compared with soy on oxidative and inflammatory stress in overweight and obese subjects. Am J Clin Nutr. 2010 Jan;91(1):16-22. doi: 10.3945/ajcn.2009.28468. Epub 2009 Nov 4. PMID 19889829
- [Derived] Zemel MB, Donnelly JE, Smith BK, Sullivan DK, Richards J, Morgan-Hanusa D, Mayo MS, Sun X, Cook-Wiens G, Bailey BW, Van Walleghen EL, Washburn RA. Effects of dairy intake on weight maintenance. Nutr Metab (Lond). 2008 Oct 24;5:28. doi: 10.1186/1743-7075-5-28. PMID 18950508